CLINICAL TRIAL: NCT04773860
Title: Muscle Energy Techniques in Chronic Obstructive Disease Patients: Effects on Pulmonary Function and Activities of Daily Living
Brief Title: Muscle Energy Techniques in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Kimberley Sevasta, Principal Investigator, University of Malta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 333797
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; METs; Muscle Energy Techniques; Dyspnoea; Activities of daily living
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with COPD
Who Masked: Participant
Masking Description: Patients shall be randomly assigned to the intervention and control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group shall be receiving a 4 week programme of Muscle Energy Techniques on the following accessory muscles; Sternocleidomastoid, Pectoralis Minor, Trapezius, Scalene muscles and Latissimus Dorsi
  Interventions: Other: Muscle Energy Techniques
- Control group (No Intervention): The control group will be taking their prescribed medication and continue with any conventional physiotherapy recommended for the individual.

INTERVENTIONS:
Other: Muscle Energy Techniques — A 4 week intervention will be carried out consisting of Muscle Energy Techniques on the accessory muscle of respiration. That is, Pectoralis Minor, Sternocleidomastoid, Upper trapezius, Scalene muscles and Latissimus Dorsi
  Arms: Experimental

SUMMARY:
Patients diagnosed with COPD as a result of hyperinflation adapt to the increased workload through shortening and overactivation of other muscles because of their dual function as muscles of the upper limb and neck motion which makes them limited in function and decreases the range of motion in these joints. Another resultant effect of these changes is the shortness of breath taking place following the inability of patients to perform daily activities.

Current research is focusing on the use of Muscle Energy Techniques (METs) for such circumstances. Therefore, this study aims to evaluate whether METs result in an improvement in rib cage mobility which could potentially lead to improvements in pulmonary function and activities of daily of living (ADLs) in a group of patients diagnosed with COPD. If positive results are obtained, such an intervention might provide a possible addition to the evidence-based interventions already available for COPD patients. The result of this intervention may provide physiotherapists with further techniques for use in such patients; ones which will be of benefit to the patients and their quality of life and also to the health services.

DETAILED DESCRIPTION:
Patients diagnosed with COPD as a result of hyperinflation adapt to the increased workload through shortening and overactivation of other muscles because of their dual function as muscles of the upper limb and neck motion which makes them limited in function and decreases the range of motion in these joints. Another resultant effect of these changes is the shortness of breath taking place following the inability of patients to perform daily activities.

Current research is focusing on the use of Muscle Energy Techniques (METs) for such circumstances. Therefore, this study aims to evaluate whether METs result in an improvement in rib cage mobility which could potentially lead to improvements in pulmonary function and activities of daily of living (ADLs) in a group of patients diagnosed with COPD. If positive results are obtained, such an intervention might provide a possible addition to the evidence-based interventions already available for COPD patients. The result of this intervention may provide physiotherapists with further techniques for use in such patients; ones which will be of benefit to the patients and their quality of life and also to the health services.

A randomised controlled trial (RCT) shall be carried out on an approximate sample of 110 patients diagnosed with COPD. Participants shall be randomly assigned to an intervention and a control group. The intervention group shall be receiving a 4 week programme of Muscle Energy Techniques whereas the control group shall continue with their prescribed medications and any conventional physiotherapy sessions suggested for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has to have been diagnosed as suffering from COPD by a medical consultant,
2. Be medically stable with no exacerbations within the past 2 months and,
3. Be between the age range of 40 to 79 years of age.

Exclusion Criteria:

1. Rheumatoid arthritis,
2. Musculoskeletal or neuromuscular pathology and,
3. Cognitive disability that could affect comprehension or execution of the intervention protocol or outcome measurements

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-02-23 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Lung function test | Week 0, Week 4 and Week 8
  Spirometry
Change in Chest expansion | Week 0, Week 4 and Week 8
  Chest expansion using a tape measure
Change in 6 Minute Walk Test | Week 0, Week 4 and Week 8
  An endurance test over a 6 minute time frame using a 30m course
Change in Manchester Related Activities of Daily Living Questionnaire | Week 0, Week 4 and Week 8
  MR-ADL is a reliable physical disability scale. It is a self-completed scale and usually takes around 10 minutes to complete. It assesses functional ability in 4 different domains, that is in the kitchen, mobility, domestic tasks and leisure activities

IPD SHARING:
Plan to Share IPD: No